CLINICAL TRIAL: NCT00103818
Title: A Double-Blind, Randomized, Multicenter, Placebo-Controlled, Parallel-Group Efficacy Study of MK0928 15 mg and 10 mg in the Treatment of Adult Outpatients With Primary Insomnia
Brief Title: An Investigational Study of MK0928 in Adult Outpatients With Insomnia (0928-014)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck Sharp & Dohme Corp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-014; MK0928-014; 2005_002
Record Dates: First submitted 2005-02-15; First posted 2005-02-16 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: gaboxadol — Duration of Treatment: 3 months
  Other Names: MK0928
Drug: Comparator: placebo (unspecified) — Duration of Treatment: 3 months

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of MK0928 for insomnia (a sleep disorder).

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients who are between the ages of 18 and 64

Exclusion Criteria:

* Adults who do not have a diagnosis of insomnia (a sleep disorder)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2005-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Patient-reported amount of sleep and time to fall asleep at night after 3 months | After 3 months

SECONDARY OUTCOMES:
Patient-reported awakenings at night | After 3 months
Sleep quality | After 3 months
Functioning after 3 months | After 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Roth T, Lines C, Vandormael K, Ceesay P, Anderson D, Snavely D. Effect of gaboxadol on patient-reported measures of sleep and waking function in patients with Primary Insomnia: results from two randomized, controlled, 3-month studies. J Clin Sleep Med. 2010 Feb 15;6(1):30-9. PMID 20191935